CLINICAL TRIAL: NCT01811394
Title: Hypofractionated Ion Irradiation (Protons or Carbon Ions) of Sacrococcygeal Chordoma
Brief Title: Ion Irradiation of Sacrococcygeal Chordoma
Acronym: ISAC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Klaus Herfarth, MD, Prof. Dr., Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISAC-01
Record Dates: First submitted 2013-03-09; First posted 2013-03-14 (Estimated); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Sacral Chordoma
Keywords: sacral chordoma; chordoma; carbon ion therapy; proton therapy; hypofractionation
MeSH Terms: conditions — Chordoma | interventions — Protons

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- protons (Experimental): 16x4GyE protons
  Interventions: Radiation: protons
- Carbon ions (Experimental): 16x4GyE carbon ions
  Interventions: Radiation: carbon ions

INTERVENTIONS:
Radiation: protons — Treatment is performed using 16 x 4 GyE protons
  Arms: protons
Radiation: carbon ions — Treatment is performed using 16 x 4 GyE carbon ions
  Arms: Carbon ions

SUMMARY:
The purpose of this study is to evaluate the safety and feasibility of primary hypofractionated irradiation of sacrococcygeal chordoma with carbon ions or protons using the raster scan technique.

DETAILED DESCRIPTION:
The primary objective of this trial is safety and feasibility of hypofractionated irradiation in patients with sacrococcygeal chordoma using protons or carbon ions in raster scan technique for primary or additive treatment after R2 resection. The evaluation is therefore based on the proportion of treatments without Grade 3-5 toxicity (CTCAE, version 4.0) up to 12 months after treatment and/or discontinuation of the treatment for any reason as primary endpoint. Local-progression free survival, overall survival and quality of life will be analyzed as secondary end points.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of sacrococcygeal chordoma
* Karnofsky performance status ≥ 70%
* Patients age 18 - 80 years
* Macroscopic tumour (MRI)
* Written informed consent

Exclusion Criteria:

* Lack of macroscopic tumour
* Tumor extension in craniocaudal direction >16cm
* Metal implants at the level of the tumor which could influence the treatment planning
* Inability of the patient to lie quiet for at least 20 minutes (eg due to pain)
* Prior radiotherapy of the pelvic region
* Simultaneous participation in another trial that could influence the results of the study
* Active medical implants without treatment approval at the time of ion irradiation (eg, cardiac pacemaker, defibrillator)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-01 (Actual); Primary Completion 2023-02 (Actual); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
safety and feasibility of hypofractionated irradiation in patients with sacrococcygeal chordoma using ions (protons or carbon ions) in raster scan technique | From date of treatment start until 12 months after treatment.
  The evaluation is based on incidence of Grade 3-5 toxicity (NCI-CTC-AE) and/or discontinuation of the treatment for any reason. Endpoint is the proportion of treatments without Grade 3-5 toxicity (NCI-CTC-AE) up to 12 months after treatment and/or discontinuation of the treatment for any reason

SECONDARY OUTCOMES:
local progression free survival (LPFS) | From date of treatment start until the date of first documented progression in MRI/CT scan assessed up to 12 months.
  local progression free survival (LPFS) is determined from start of treatment until local progression in imaging (>10% size increase)
Overall survival (OS) | From date of treatment start until the date of death from any cause assessed up to 12 months.
  Further objectives are overall survival (OS) from date of treatment start until the date of death from any cause assessed up to 12 months
Quality of life (QoL) | From date of treatment start up to 12 months. Evaluation at treatment start, at the end of treatment and 12 months after treatment.
  Quality of life (QoL) evaluated with EORTC-QLQ30 questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Heidelberg, Radiooncology, HIT, Heidelberg, Germany

REFERENCES:
- [Background] Uhl M, Edler L, Jensen AD, Habl G, Oelmann J, Roder F, Jackel O, Debus J, Herfarth K. Randomized phase II trial of hypofractionated proton versus carbon ion radiation therapy in patients with sacrococcygeal chordoma-the ISAC trial protocol. Radiat Oncol. 2014 Apr 29;9:100. doi: 10.1186/1748-717X-9-100. PMID 24774721